CLINICAL TRIAL: NCT02957942
Title: Repetitive Transcranial Magnetic Stimulation in Spasmodic Dysphonia
Brief Title: rTMS in Spasmodic Dysphonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PSYCH-2016-25008
Record Dates: First submitted 2016-10-26; First posted 2016-11-08 (Estimated); Results first posted 2020-10-01 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Spasmodic Dysphonia; Laryngeal Dystonia
Keywords: Repetitive transcranial magnetic stimulation (rTMS); Spasmodic dysphonia; Dystonia
MeSH Terms: conditions — Dysphonia; Dystonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Spasmodic Dysphonia (Experimental): 1Hz repetitive transcranial magnetic stimulation (rTMS)
  Interventions: Device: 1Hz repetitive transcranial magnetic stimulation (rTMS)
- Healthy control (Active Comparator): Healthy adults 1Hz repetitive transcranial magnetic stimulation (rTMS)
  Interventions: Device: 1Hz repetitive transcranial magnetic stimulation (rTMS)

INTERVENTIONS:
Device: 1Hz repetitive transcranial magnetic stimulation (rTMS) — 1 session of low-frequency rTMS (1Hz, 1200 pulses, 20 minutes)

SUMMARY:
Focal dystonia is a neurological movement disorder characterized by excessive involuntary muscle contractions of any body part. Spasmodic dysphonia (SD) is a type of focal dystonia characterized by excessive contraction of intrinsic muscles in the larynx, leading to difficulty in speaking and affecting effective communication. The cause of SD is unknown and there are no treatments that produce long-term benefits. Previous studies have suggested that SD and other focal dystonias are associated with decreased inhibition in sensorimotor areas in the brain. However, no studies have investigated the effects of modulating excitability of the laryngeal motor cortex in healthy individuals or SD. The goal of this pilot project is to determine if brain excitability of the laryngeal motor cortex can be changed with low-frequency inhibitory repetitive transcranial magnetic stimulation (rTMS) in individuals with SD and healthy controls. Considering that rTMS at low frequencies (≤1 Hz) produces lasting inhibition in the brain, and that SD is associated with decreased cortical inhibition, the purpose of this pilot study is to determine safety, feasibility and response to 1Hz rTMS to the laryngeal motor cortex in individuals with SD and healthy people. The results will help understand changes associated with the disorder, as well as contribute to the development of future clinical interventions for SD.

ELIGIBILITY:
Inclusion Criteria:

* Primary inclusion for spasmodic dysphonia:

  1. Diagnosis of adductor spasmodic dysphonia
  2. Symptoms at worst severity if receiving regular botulinum injections
* Primary inclusion for healthy participants (controls):

  1. Absence of vocal fold pathology

Exclusion Criteria:

* Primary exclusion for participants with spasmodic dysphonia:

  1. Other forms of dystonia
  2. Vocal fold pathology or paralysis
  3. Diagnosis of voice tremor
  4. Laryngeal surgery
  5. Laryngeal cancer or neurological condition other than dystonia
  6. Contraindication to TMS
  7. Medications with effect on central nervous system
  8. Inability to complete tasks associated with study
  9. Adult lacking ability to consent
* Primary exclusion for healthy participants (controls):

  1. Any health condition or disability that would interfere with participation
  2. Contraindications to TMS
  3. Medications with effect on central nervous system
  4. Adult lacking ability to consent

TMS contraindications:

* The only absolute contraindication to TMS/rTMS is the presence of metallic hardware in close contact to the discharging coil (such as cochlear implants, deep brain stimulator, or medication pumps). In such instances there is a risk of inducing malfunctioning of the implanted devices.
* Conditions classified as of increased or uncertain risk are listed below (Rossi et al., 2009; Rossini et al., 2015). Persons under those circumstances will be excluded from the study.

  1. Pregnancy
  2. Bipolar disorder
  3. Epilepsy or history of seizure episodes in the past two years
  4. Vascular, traumatic, tumoral, infectious, or metabolic lesion of the brain, even without history of seizure, and without anticonvulsant medication
  5. Use of medications that potentially lower seizure threshold
  6. Severe or recent heart disease

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mo Chen, PhD, Principal Investigator — University of Minnesota; Teresa J Kimberley, PhD, PT, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Noninvasive Neuromodulation Laboratory, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Background] Rossini PM, Burke D, Chen R, Cohen LG, Daskalakis Z, Di Iorio R, Di Lazzaro V, Ferreri F, Fitzgerald PB, George MS, Hallett M, Lefaucheur JP, Langguth B, Matsumoto H, Miniussi C, Nitsche MA, Pascual-Leone A, Paulus W, Rossi S, Rothwell JC, Siebner HR, Ugawa Y, Walsh V, Ziemann U. Non-invasive electrical and magnetic stimulation of the brain, spinal cord, roots and peripheral nerves: Basic principles and procedures for routine clinical and research application. An updated report from an I.F.C.N. Committee. Clin Neurophysiol. 2015 Jun;126(6):1071-1107. doi: 10.1016/j.clinph.2015.02.001. Epub 2015 Feb 10. PMID 25797650
- [Background] Summers RL, Chen M, Kimberley TJ. Corticospinal excitability measurements using transcranial magnetic stimulation are valid with intramuscular electromyography. PLoS One. 2017 Feb 23;12(2):e0172152. doi: 10.1371/journal.pone.0172152. eCollection 2017. PMID 28231250
- [Background] Kimberley TJ, Schmidt RL, Chen M, Dykstra DD, Buetefisch CM. Mixed effectiveness of rTMS and retraining in the treatment of focal hand dystonia. Front Hum Neurosci. 2015 Jul 9;9:385. doi: 10.3389/fnhum.2015.00385. eCollection 2015. PMID 26217209
- [Background] Chen M, Summers RL, Goding GS, Samargia S, Ludlow CL, Prudente CN, Kimberley TJ. Evaluation of the Cortical Silent Period of the Laryngeal Motor Cortex in Healthy Individuals. Front Neurosci. 2017 Mar 7;11:88. doi: 10.3389/fnins.2017.00088. eCollection 2017. PMID 28326007
- [Derived] Prudente CN, Chen M, Stipancic KL, Marks KL, Samargia-Grivette S, Goding GS, Green JR, Kimberley TJ. Effects of low-frequency repetitive transcranial magnetic stimulation in adductor laryngeal dystonia: a safety, feasibility, and pilot study. Exp Brain Res. 2022 Feb;240(2):561-574. doi: 10.1007/s00221-021-06277-4. Epub 2021 Dec 2. PMID 34859288

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Spasmodic Dysphonia | Healthy Control
Started | 7 | 13 (7 healthy individuals were recruited as control; 6 were recruited for practicing experiment details.)
Completed | 7 | 6
Not Completed | 0 | 7
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Practicing experiment protocol | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Spasmodic Dysphonia | Healthy Control | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 13
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (3.8) | 53.2 (6.6) | 57.4 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 7 | 5 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Adverse Response to rTMS
Description: Count of participants who experience and adverse response to rTMS treatment.
Time Frame: 2.5 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Spasmodic Dysphonia | Healthy Control
Number analyzed (Participants) | 7 | 6
Participants | 0 | 0

2. Primary Outcome: Change in Duration of Cortical Silent Period (CSP)
Description: The change from baseline in CSP duration will be reported. The CSP is an interruption of voluntary muscle contraction after single pulse transcranial stimulation. The duration of the period of silent muscle activity will be measured to test the effects of rTMS intervention. There is no known clinical relevance for this outcome measure.
Time Frame: baseline and 2.5 hours
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Spasmodic Dysphonia | Healthy Control
Number analyzed (Participants) | 7 | 6
milliseconds | -2.4 (10.6) | 3.6 (8.8)

3. Secondary Outcome: Change in Number of Voice Breaks
Description: Changes from baseline in the number of voice breaks during speech will be reported. Voice breaks will be measured by asking subjects to repeat 10 sentences. The frequency of voice breaks in the recorded 10 sentences will be counted.
Time Frame: baseline and 2.5 hours
Measure: Mean (Standard Deviation); unit: total voice breaks
Arm/Group | Spasmodic Dysphonia | Healthy Control
Number analyzed (Participants) | 7 | 6
total voice breaks | -1.3 (4.7) | 0 (0)

4. Secondary Outcome: Change in Voice Quality (Overall Severity) With the Consensus Auditory-Perceptual Evaluation of Voice (CAPE-V)
Description: CAPE-V (overall severity) testing before and after rTMS consisted of the repetition of six sentences and two sustained vowels (/a/;/i/). A short sample of spontaneous speech (approximately 60s) was also collected for qualitative analysis of voice. The CAPE-V ratings were completed by three assessors who were blinded to group and pre/post-test. The assessors listened to the voice recordings for each participant and rated them for all six parameters listed above from 0 to 100, with higher values indicating worse severity. Ratings for each voice parameter were then averaged across the three assessors. We chose to analyze the change in the CAPE-V parameter for "Overall Severity" to represent an overall assessment of voice quality from pre- to post-rTMS (Post Score - Pre Score) as it had the greatest likelihood of detecting any small changes that may be perceived.
Time Frame: baseline and 2.5 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Spasmodic Dysphonia | Healthy Control
Number analyzed (Participants) | 7 | 6
score on a scale | -3.7 (10.5) | 0.9 (5.2)

5. Secondary Outcome: Change in Cepstral Peak Prominence Smoothed (CPPS)
Description: Quantitative assessment of voice quality was completed with acoustic analysis of each participant's production of the ten sentences from the Spasmodic Dysphonia Attribute Inventory (SDAI). A custom script in Praat (Boersma & Weenink, 2018) was used to calculate cepstral peak prominence smoothed (CPPS) for each sentence production. CPPS is a relatively new measure that reflects vocal fold periodicity and noise components in the vocal spectrum. CPPS has been found to be correlated with perceived severity of voice symptoms and higher CPPS values represent a more normal vocal quality. CPPS values (in dB) were averaged across the ten sentences of the SDAI to derive an average CPPS for each participant before and after rTMS. Change for each participant was calculated as the average CPPS at post-rTMS minus average CPPS at pre-rTMS. The values for each group were then averaged to report the average change in CPPS for Controls and Spasmodic Dysphonia.
Time Frame: baseline and 2.5 hours
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Spasmodic Dysphonia | Healthy Control
Number analyzed (Participants) | 7 | 6
dB | 0.1 (0.7) | 0.3 (0.8)

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Spasmodic Dysphonia | Healthy Control
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 7/7 | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Spasmodic Dysphonia (N=7) | Healthy Control (N=6)
Throat Pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Tenderness on Skin Area of Insertion (Injury, poisoning and procedural complications) | 3 (3) | 5 (5)
Neck Pain (General disorders) | 1 (1) | 4 (4)
Dental Pain/Discomfort (General disorders) | 0 (0) | 1 (1)
Dizziness (General disorders) | 0 (0) | 1 (1)
Other(fatigue) (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-02): https://cdn.clinicaltrials.gov/large-docs/42/NCT02957942/Prot_SAP_000.pdf